# Prediction of spontaneous preterm birth in multiple gestation by cervical elastogram

# **Investigators:**

LEUNG Tak Yeung
HUI Shuk Yi Annie
POON Liona Chiu Yee
LU Jing
CHENG Yvonne Kwun Yue

# **Affiliation:**

Department of Obstetrics and Gynaecology, The Chinese University of Hong Kong, Prince of Wales Hospital

Compliance with the Declaration of Helsinki: Yes

Protocol version: 1.3 (dated 18 Apr 2018)

### **Background**

Preterm birth is the leading cause of perinatal morbidity and mortality in multiple pregnancy, and the medical and educational expenditure and lost productivity associated with preterm birth is very high.

The risk of preterm delivery in singleton pregnancy is 5-7%, and that in twin pregnancy is 7-8 fold higher than singleton pregnancy. [1] Identification of pregnant women at risk of preterm birth could allow intervention to reduce their risk. Treatment such as progesterone, cervical pessary, and surgical cerclage in selected cases have been shown to be effective measures to reduce the risk of preterm delivery in singletons. [2-4] Prevention of preterm birth in multiple pregnancy is more challenging. A lot of preventive methods studied, including bed rest, tocolysis, nutritional adjustment, cerclage and cervical pessary, have not been shown to be effective. [5-10] Until very recently, a study have found that vaginal progesterone is effective in reducing preterm birth < 33 weeks in twin pregnancy with a risk reduction of 30%, and a significant reduction in neonatal death, respiratory distress syndrome, and composite morbidity and mortality was also demonstrated. [11]

Premature dilatation and shortening of cervix have been demonstrated to be a very good predictor of preterm birth in singleton as well as twin pregnancies. [12-25] The ability to identify pregnant women with short cervix allows timely intervention to reduce their risk. Nevertheless, not all women who end up having preterm birth have a short cervix, prompting identification of other cervical signs to increase the prediction of preterm birth.

Recently, a new ultrasound technology called sonoelastograhy has enabled the measurement of tissue stiffness. [26,27] It has been widely applied in assessment of breast lump and liver cirrhosis, as the tissue is stiffer in case of malignancy and cirrhosis. [28,29] Sonoelastography is potentially useful for the objective assessment of cervical consistency which could be related to risk of preterm birth. A recent study has shown that strain in the internal cervical os has been shown to be associated with spontaneous preterm delivery in singleton pregnancies. [30] This study has shown some promising results in the use of elastography in prediction of preterm delivery, however, it is limited by the fact that the sonographic technique used is strain elastography, which could be affected by the pressure of the probe on the cervix. On the other hand, shear wave elastography creates images based on moving waves and is

therefore a dynamic technique to assess energy loss when it travels through tissue. The benefit being that the results are relatively independent of the operator, because strain elastography would not be affected by the pressure exerted on the cervix. Furthermore, although strain elastography is good for measuring stiffness differences, such as stiff tumour inside softer liver tissue, it is not designed to measure overall variations in stiffness, as in cervical consistency. [31]

The aim of this study is to assess the cervical consistency by shear wave elastography in prediction of preterm birth in multiple pregnancies.

### Hypothesis:

We hypothesize that a 'soft' cervix as indicated by shear wave elastography is positively associated with the risk of preterm birth in twin pregnancies.

# **Design of study**

This is a prospective non-interventional observational study.

#### Methods

Chinese women carrying multiple pregnancies attending antenatal visit at Prince of Wales Hospital are invited to join the study. The study details will be explained by the research assistant or one of the investigators and informed consent will be obtained. Demographic data, antenatal history will be obtained. Exclusion criteria include an age of less than 18 years, non-Chinese, inability to provide consent and those who refuse to join.

Other risk factors of preterm delivery will also be documented:

- known cervical insufficiency
- surgical cerclage or pessary in previous pregnancy
- history of preterm prelabour rupture of membranes (PPROM) or spontaneous preterm birth before 34 weeks
- history of cervical surgery including cone biopsy, loop electrosurgical excision procedure, cervical tear repair, etc

- short cervix <2.5cm cervical length
- painless cervical os dilatation

A trained researcher or an obstetrician will perform transvaginal scan for the cervix on the same day of the antenatal visit, or on a separate study date, if necessary. Measurements will be done at 5 visits: 11-15 weeks, 16-19 weeks, 20-23 weeks, 24-27 weeks, 28-32 weeks. The number of visits will be depended on when the subjects are initially recruited.

The following will be measured:

- Cervical consistency by sonoelastogrpahy
- Cervical length by 2D ultrasonography
- Posterior cervical angle by 2D ultrasonography
- Fetal viability

The TVS measurement of the cervical length, posterior angle and sonoelastography is elaborated as follow:

- An USG machine equipped with shear wave elastography (SWE) is used (scale set to 0-100kPa)
- Participants are asked to empty the urinary bladder before TVS, and lie in lithotomy position
- A 12-3MHz transvaginal transducer (with double condom cover and lubricant) is inserted into the vagina gently, with no pressure exerted on the cervix
- The mid-sagittal view of the cervix is obtained and magnified
- The cervical length and the posterior angle are then measured as described in our previous study [32, 33]
- SWE mode is then switched on and a color box showing the elastogram is demonstrated
- The color box will be placed at the central part of the anterior lip of the cervix (more proximal to the USG probe than the posterior lip)
- Once the color box is uniformly filled with color signals on the elastogram, the image is frozen and a region of interest (Q-box) of size 10mm is placed to measure the tissue elasticity (in term of kPa).
- Women will be asked to perform Valsalva maneuvers and mesurements of cervical

length, posterior angle and elastography will be obtained under such maneuver.

- The acquisition time is kept short within ten seconds to avoid erroneous data collection.
- Images will be saved for future analyses, if necessary.

Women, including those who are found to have a short cervix, will be managed according to the departmental protocol and their obstetric management will not be affected by the study. The obstetrician will be blinded to the finding of the sonoelastography and the finding would not affect the obstetric management of the women.

The delivery data and neonatal outcome will be collected from the medical notes and hospital electronic system before the women are discharged after their delivery.

#### Main outcome measures:

- 1. The association of cervical consistency in mid trimester with spontaneous preterm birth in women carrying multiple pregnancies.
- 2. The change in cervical consistency during pregnancy in women carrying multiple pregnancies.

## **Sample Size:**

The risk of preterm birth <34 weeks in twin pregnancies is approximately 20%. A sample size of 120 was determined as being sufficient to test the diagnostic performance of cervical elasticity in mid trimester assuming that the risk of preterm delivery <34 weeks vs >34 weeks is 1:5 and that cervical elasticity area under curve (AUC) of the receiver operating characteristics (ROC) curve was 0.7, with 80% power and alpha of 5%. From the start of recruitment up to March 2018, only 15 (34.1%) out of 44 cases had completed all five serial cervix measurements. We aim to collect 120 completed set of measurements to allow our result to be statistically significant. Therefore, we increase the sample size to 200.

# **Statistical Analysis:**

Changes in the cervical elastography will be compared using the Student paired two-tailed t test, and in the case of unequal standard deviation (SD), using a Wilcoxon signed-rank paired

two-tailed test. For comparison of frequencies, Chi-square test, or a two-sided Fisher exact test will be used where appropriate. Linear regression will be used to assess the correlations. Statistical analysis was performed using the Statistical Package for Social Science (SPSS) version 20.0 (SPSS, IL). The level of statistical significance is set at p<0.05 (two-sided).

## **Purpose and Potential**

A significant improvement in the prediction of preterm delivery allows accurate differentiation of those women who would benefit from treatment for prevention of preterm birth in multiple pregnancy. This would avoid unnecessary intervention, reduce maternal and fetal complications, and has a potential to save medical cost.

### **Key References**

- 1. Hamilton BE, Martin JA, Osterman MJ, Curtin SC, Matthews TJ. Births: Final Data for 2014. Natl Vital Stat Rep 2015;64:1-64.
- Dodd JM, Jones L, Flenady V, Cincotta R, Crowther CA. Prenatal administration of progesterone for preventing preterm birth in women considered to be at risk of preterm birth. Cochrane Database Syst Rev 2013; 7: CD004947.
- 3. Goya M, Pratcorona L, Merced C, et al. Cervical pessary in pregnant women with a short cervix (PECEP): an open-label randomised controlled trial. Lancet 2012;379:1800-6.
- 4. Sanchez-Ramos L, Kaunitz AM, Delke I. Progestational agents to prevent preterm birth: a meta-analysis of randomized controlled trials. Obstet Gynecol 2005; 105:273–279.
- 5. Crowther CA, Han S. Hospitalisation and bed rest for multiple pregnancy. Cochrane Database Syst Rev 2010;7:CD000110.
- 6. Yamasmit W, Chaithongwongwatthana S, Tolosa JE, Limpongsanurak S, Pereira L, Lumbiganon P. Prophylactic oral betamimetics for reducing preterm birth in women with a twin pregnancy. Cochrane Database Syst Rev 2015;12:CD004733.
- 7. Goodnight W, Newman R; Society of Maternal-Fetal Medicine. Optimal nutrition for improved twin pregnancy outcome. Obstet Gynecol 2009;114:1121-1134.
- 8. Rafael TJ, Berghella V, Alfirevic Z. Cervical stitch (cerclage) for preventing preterm birth in multiple pregnancy. Cochrane Database Syst Rev 2014;9:CD009166.
- 9. Liem S, Schuit E, Hegeman M, Bais J, de Boer K, Bloemenkamp K, et al. Cervical pessaries for prevention of preterm birth in women with a multiple pregnancy (ProTWIN): a multicenter, open-label randomized controlled trial. Lancet 2013;382:13411349.
- 10. Nicolaides KH, Syngelaki A, Poon LC, de Paco Matallana C, Plasencia W, Molina FS, et al. Cervical pessary placement for prevention of preterm birth in unselected twin pregnancies: a randomized controlled trial. Am J Obstet Gynecol 2016;214:3.e1-9.

- 11. Romero R, Conde-Agudelo A, El-Refaie W, Rode I, Brizot ML, Cetingoz E, et al. Vaginal progesterone decreases preterm birth and neonatal morbidity and mortality in women with a twin gestation and a short cervix: an updated meta-analysis of individual patient data. Ultrasound Obstet Gynecol. 2017;49:303-314.
- 12. Anderson HF, Nugent CE, Wanty SD, Hayashi RH. Prediction of risk of preterm delivery by ultrasonographic measurement of cervical length. Am J Obstet Gynecol 1990;163:859-67.
- 13. Iams JD, Goldenberg RL, Meis PJ, Mercer BM, Moawad A, Das A, et al. The length of the cervix and the risk of spontaneous premature delivery. National Institute of Child Health and Human Development Maternal Fetal Medicine Unit Network. N Engl J Med 1996;334:567-72.
- 14. Heath VC, Southall TR, Souka AP, Elisseou A, Nicolaides KH. Cervical length at 23 weeks of gestation: prediction of spontaneous preterm delivery. Ultrasound Obstet Gynecol 1998;12:312-7.
- 15. Welsh A, Nicolaides K. Cervical screening for preterm delivery. Curr Opin Obstet Gynecol 2002;14:195-202.
- 16. Hassan S, Romero R, Hendler I, Gomez R, Khalek N, Espinoza J, et al. A sonographic short cervix as the only clinical manifestation of intra-amniotic infection. J Perinat Med 2006;34:13-9.
- 17. Hassan SS, Romero R, Berry SM, Dang K, Blackwell SC, Treadwell MC, et al. Patients with an ultrasonographic cervical length < or =15mm have nearly a 50% risk of early spontaneous preterm delivery. Am J Obstet Gynecol 2000;182:1458-67.
- 18. Romero R. Prevention of spontaneous preterm birth: the role of sonographic cervical length in identifying patients who may benefit from progesterone treatment. Ultrasound Obstet Gynecol 2007;30:675-86.
- 19. Crane JM, Hutchens D. Transvaginal sonographic measurement of cervical length to predict preterm birth in asymptomatic women at increased risk: a systematic review. Ultrasound Obstet Gynecol 2008;31:579-87.
- 20. Vaisbuch E, Romero R, Erez O, Kusanovic JP, Mazaki-Tovi S, Gotsch F, et al. Clinical significance of early (<20 weeks) vs. late (20-24 weeks) detection of sonographic short cervix in asymptomatic women in the mid-trimester. Ultrasound Obstet Gynecol 2010;36:471-81.
- 21. Barros-Silva J, Pedrosa AC, Matias A. Sonographic measurement of cervical length as a predictor of preterm delivery: a systematic review. J Perinat Med 2014;42:281-93.
- 22. Melamed N, Pittini A, Hiersch L, Yogev Y, Korzeniewski SJ, Romero R, Barrett J. Do serial measurements of cervical length improve the prediction of preterm birth in asymptomatic women with twin gestations? Am J Obstet Gynecol 2016;215(5):616.e1-616.e14.
- 23. Melamed N, Pittini A, Hiersch L, Yogev Y, Korzeniewski SS, Romero R, Barrett J. Serial cervical length determination in twin pregnancies reveals 4 distinct patterns with prognostic significance for preterm birth. Am J Obstet Gynecol 2016;215(4):476.e1-476.e11.

- 24. El-Gharib MN, Albehoty SB. Transvaginal cervical length measurement at 22- to 26-week pregnancy in prediction of preterm births in twin pregnancies. J Matern Fetal Neonatal Med 2017;30(6):729-732.
- 25. Kindinger LM, Poon LC, Cacciatore S, MacIntyre DA, Fox NS, Schuit E, Mol BW, Liem S, Lim AC, Serra V, Perales A, Hermans F, Darzi A, Bennett P, Nicolaides KH, Teoh TG. The effect of gestational age and cervical length measurements in the prediction of spontaneous preterm birth in twin pregnancies: an individual patient level meta-analysis. BJOG. 2016;123(6):877-84.
- 26. Bercoff J, Tanter M, Fink M. Supersonic shear imaging: a new technique for soft tissue elasticity mapping. IEEE Trans Ultrason Ferroelectr Freq Control. 2004;51(4):396-409.
- 27. Ophir J, Cespedes I, Ponnekanti H, Yazdi Y, Li X. Elastography: a quantitative method for imaging the elasticity of biological tissues. Ultrason Imaging 1991;13:111-34.
- 28. Berg WA, Cosgrove DO, Doré CJ, Schäfer FK, Svensson WE, Hooley RJ, Ohlinger R, Mendelson EB, Balu-Maestro C, Locatelli M, Tourasse C, Cavanaugh BC, Juhan V, Stavros AT, Tardivon A, Gay J, Henry JP, Cohen-Bacrie C, and the BE1 Investigators. Shear-wave elastography improves the specificity of breast US: the BE1 multinational study of 939 masses. Radiology 2012;262(2):435-49.
- 29. Bavu E, Gennisson JL, Couade M, Bercoff J, Mallet V, Fink M, Badel A, Vallet-Pichard A, Nalpas B, Tanter M, Pol S. Noninvasive in vivo liver fibrosis evaluation using supersonic shear imaging: a clinical study on 113 hepatitis C virus patients. Ultrasound Med Biol 2011;37:1361-73.
- 30. Hernandez-Andrade E, Garcia M, Ahn H, Korzeniewski SJ, Saker H, Yeo L, et al. Strain at the internal cervical os assessed with quasi-static elastography is associated with the risk of spontaneous preterm delivery at <=34 weeks of gestation. J Perinat med 2015;43(6):657-666.
- 31. Fruscalzo A, Mazza E, Feltovich H, Schmitz R. Cervical elastography during pregnancy: a critical review of current approaches with a focus on controversies and limitations. J med Ultrasonics 2016;43:493-504.
- 32. Cheung CW, Leung TY, Sahota DS, Chan OK, Chan LW, Fung TY, Lau TK. Outcome of induction of labour using maternal characteristics, ultrasound assessment and biochemical state of the cervix. J Matern Fetal Neonatal Med 2010;23(12):1406-12.
- 33. Kolkman DG, Verhoeven CJ, Brinkhorst SJ, van der Post JA, Pajkrt E, Opmeer BC, Mol BW. The Bishop score as a predictor of labor induction success: a systematic review. Amer J Perinatol 2013;30(8):625-30.